CLINICAL TRIAL: NCT03666650
Title: Relationship of Edoxaban Plamsa Concentration and Blood Coagulation in Healthy Volunteers Using Standard Laboratory Tests and Viscoelastic Analysis
Brief Title: NOAC Plasma Concentration and Blood Coagulation in Healthy Volunteers
Acronym: EdoRot
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Marko Peltoniemi, MD, PhD, Study Principal Investigator, Perioperative Services, Intensive Care and Pain Therapy, Turku University Hospital, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: T224/2018
Record Dates: First submitted 2018-09-08; First posted 2018-09-12 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Blood Coagulation Disorder
MeSH Terms: conditions — Blood Coagulation Disorders | interventions — edoxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rotem (Other)
  Interventions: Drug: Edoxaban 60 MG

INTERVENTIONS:
Drug: Edoxaban 60 MG — Viscoelastic analysis and standard laboratory tests after edoxaban ingestion

SUMMARY:
Relationship of edoxaban plasma concentration and blood coagulation in healthy volunteers using standard laboratory tests and viscoelastic analysis

ELIGIBILITY:
Inclusion Criteria:

healthy

Exclusion Criteria:

intolerance of the study drug history of bleeding disorder or similar

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
correlation of edoxaban peak plasma concentrations and viscoelastic analysis | 1 day
  viscoelastic test values and blood coagulation laboratory parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Southwest Finland, Finland

IPD SHARING:
Plan to Share IPD: No